CLINICAL TRIAL: NCT06071663
Title: Clinical and Radiographic Evaluation of Single-Versus Two-visit Pulpectomy in Primary Molars: Randomized Controlled Clinical Trial
Brief Title: Single and Two-visit Pulpectomy in Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Moustafa Reda, Sherbin/Dakhlia/Egypt, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: A0603023PP
Record Dates: First submitted 2023-10-01; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Dental Pulp Necroses
Keywords: Pulpectomy, single visit, two visits
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single visit (Active Comparator): Necrotic primary molar treated in single visit
  Interventions: Procedure: Single and two visits pulpectomy
- Two visits (Active Comparator): Necrotic primary molar treated in two visits
  Interventions: Procedure: Single and two visits pulpectomy

INTERVENTIONS:
Procedure: Single and two visits pulpectomy — Comparison of clinical and radiographic outcome of Single and two visits pulpectomy

SUMMARY:
A total of 64 primary molars of 5-8 years old children will be randomly selected from Pediatric dental clinic at Faculty of Dentistry, Mansoura University.

Children will have two bilateral carious primary molars indicated for pulpectomy ; One side will be treated in one visit and the other will be treated in two visits.

Clinical and radiographic evaluation for 3 , 6, 12 months

DETAILED DESCRIPTION:
All the pulpectomy steps will be carried out by a single operator. After confirming the diagnosis clinically and radiographically, the necrotic tooth will be anesthetized by local anesthesia and isolated by rubber dam.

Caries will be removed by sterile round diamond burs. Proper access cavity will be prepared with complete deroofing and the pulp chamber will be irrigated by saline 0.9%. The working length will be established by apex locator and confirmed by periapical film (1 mm short of radiographic apex). Mechanical instrumentation will be done using rotary files followed by irrigation with no excessive pressure between files using sodium hypochlorite 2.5%. Then, root canal system will be dried by sterile paper points.

In case of single visit pulpectomy (21):

Root canals will be obturated by metapex and the tooth will be finally restored by glass ionomer filling and stainless-steel crown.

In case of two visit pulpectomy (13):

First, root canals will be filled by calcium hydroxide powder mixed with saline followed by temporary coronal restoration and left for 7 days.

In the second visit, calcium hydroxide will be removed from the canals using K -files then irrigated by NaOCL 2.5%. The canals will be dried by sterile paper points before obturation and final restoration as mentioned in single- visit treatment protocol. A postoperative periapical x-ray film will be taken for future review.

Clinical and radiographic follow up will be carried out after 3, 6, 12 months respectively.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative 5-8 years old children with no systemic diseases or chronic conditions. _Every child should have bilateral necrotic primary molars indicated for pulpectomy with sufficient coronal tooth structure.

Exclusion Criteria:

* Children received antibiotics in the past month before the study. Primary molars with sinus tract, abscess, or facial cellulitis. Primary molas with root resorption exceeding one third of root length

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2023-10-05 (Estimated); Primary Completion 2024-01-05 (Estimated); Study Completion 2024-10-05 (Estimated)

PRIMARY OUTCOMES:
Clinical and Radiographic outcomes | 3 , 6 and 12 months
  Proportion of clinical and radiographic success in both treatment protocols

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Moustafa Fareag, Professor, Study Director — Pediatric dentistry department. MANSOURA UNIVERSITY